CLINICAL TRIAL: NCT00891969
Title: The Process and Outcomes of Treatment Decision-Making Communication Between Oncologists and Newly Diagnosed Female Breast-Cancer Patients
Brief Title: Treatment Decision Making Between Oncologists and Women With Newly Diagnosed Breast Cancer and Their Healthy Companions
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 040810; P30CA072720 (NIH); 0220080300
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RATIONALE: A study that looks at communication between patients and doctors may help oncologists improve patient satisfaction with their treatment plan.

PURPOSE: This phase I trial is studying treatment decision making between oncologists and women with newly diagnosed breast cancer and their healthy companions.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the association between women's and physicians' participatory communication behaviors (e.g., patients asking questions, physicians soliciting questions) on treatment decision-making process and health outcomes.

Secondary

* To capture the language used in the treatment-decision interactions.
* To assess the degree of variation in the language used among physicians and patients who are active participants and those who are less inclined to participate in the treatment decision-making interaction.

OUTLINE: Patients and their companions undergo consultation with the physician for treatment decision making. The treatment discussion is audio/videotaped for approximately 45 minutes.

Patients complete one short survey prior to physician consultation. After the treatment discussion, patients complete two short surveys, one immediately after the visit in the waiting room before leaving for the day, and the second one a week after the visit by a web-based survey or by mail.

PROJECTED ACCRUAL: A total of 300 women with breast cancer and 600 companions of these women will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Woman with newly diagnosed early-stage breast cancer
  * Caregiver or companion willing to participate in study

PATIENT CHARACTERISTICS:

* Speaks native English or has learned to speak English fluently
* Patient's companion ≥ 18 years old (if applicable)
* Able to complete questionnaires without assistance
* Not pregnant

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, early-stage, female, breast-cancer patients who are scheduled to see a participating surgical oncologist for an initial treatment decision making visit
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The association between patients' and physicians' participatory communication and psychosocial outcomes. | Pre- and post-Initial treatment decision making visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Kearney, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States